CLINICAL TRIAL: NCT03131284
Title: Prevention of Obesity in Toddlers (PROBIT): a Randomized Clinical Trial of Primary Pediatric Care From Birth Onwards.
Brief Title: Prevention of Obesity in Toddlers (PROBIT) Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, Claudio Maffeis, Professor, Azienda Ospedaliera Universitaria Integrata Verona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 368 CEP
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Families of newborns whose paediatrician is assigned to the control arm, receive usual education about nutrition and lifestyle, during their child's first two years of life.
- Intensive education. (Experimental): Families of newborns whose paediatrician is assigned to the intervention arm, receive standardized lifestyle counseling along with educational written material about their child's first two years of life, which corresponds to the experimental treatment.
  Interventions: Behavioral: Intensive education

INTERVENTIONS:
Behavioral: Intensive education — For each well visit within the first two years of their child's life, parents are provided with oral and written information on behaviors to adopt for their child to be protected from obesity: breast feeding, feeding on demand, responsive feeding, correct time of introduction of complementary feeding, portions shaped on the child's appetite, avoiding "pressing the child to eat more" and rewarding or punishing the child with food, avoiding added sugar and beverages other than milk and water, practicing active game with the child, alternating protein sources correctly and avoiding protein excess. Written menus examples and coloured photos of average portions are given for complementary feeding. Parents are also provided with information about health consequences of childhood obesity.
  Arms: Intensive education.

SUMMARY:
AIM:

to reduce the prevalence of overweight and obesity at two years of age in the intervention group compared to the control group.

METHODS:

Eleven primary paediatricians were randomized to the intervention group and intensively trained about the trial intervention. Each of them was asked to consecutively recruit the parents of at least 30 newborns taken in charge within the first six months of the study, and to provide them with standardized oral and written information on protective practices during all the well visits scheduled in the first two years of the child's life.

Another eleven primary paediatricians were randomized to the control group, and were asked to consecutively recruit the parents of at least 30 newborns taken in charge within the first six months of the study and to provide them with usual care and follow-up. When all recruited children have completed the second year of life, the two groups of toddlers will be compared as regards the prevalence of overweight/obesity, defined by WHO cut-offs of the weight/length ratio.

DETAILED DESCRIPTION:
INTRODUCTION:

Childhood overweight and obesity represent a serious public health emergency for most western and westernized countries. In fact, obesity prevalence has been increasing for several decades in these countries and weight excess is associated with severe psychological and physical complications, such as depression, diabetes, infertility and cardiovascular disease. As a consequence, childhood obesity is associated with a significant increase of the risk of premature death from endogenous causes. In the Northern Italy, the overall prevalence of overweight/obesity among school children is 25 to 33%, among the highest in Europe.

Childhood overweight and obesity are chronic diseases, with low rate of resolution either spontaneous or following medical care, and with high rates of persistence into adulthood as well as worsening and/or relapse after temporary improvements. Thus, prevention is recognized as the most promising strategy to combat the obesity epidemic during childhood.

The meta-analysis of pediatric prevention trials has highlighted a poor effectiveness of interventions targeting school children and a scarcity of data on interventions targeting the infancy. This is internationally recognized as an important gap of the state of the art on obesity prevention. In fact, the mechanisms leading to obesity may be triggered, in most children, during the first months or years of life, making preventive interventions too late and non effective for several children who are already overweight or obese at three years of age. The few existing prevention trials targeting pre-school children have been more encouraging than those concerning school-age, especially when considering interventions based on the education of parents rather than on modifications of extra-family environment (kinder-garden, etc…).

There are several known modifiable risk factors for early growth acceleration, which may inspire potentially effective interventions to prevent overweight and obesity in toddlers. These risk factors concern breast feeding, complementary feeding, nutrition during the first and second year of life, parenting style, feeding practices (i.e. scheduled feeding, responsive feeding, feeding to calm, etc…), and overall lifestyle (active play and sleeping patterns).

The PROBIT trial aims to decrease the prevalence of overweight/obesity at two years of life, in a group of toddlers whose parents are provided with an intensive standardized educational intervention from their child' s birth onwards (intervention arm), compared to a group of toddlers whose parents are not provided with any additional intervention besides the usual care and follow-up provided by their paediatrician (control arm).

The secondary aims of the trial are:

* to improve the feeding practices during the first two years of life in the intervention group compared to the control group;
* to reduce the prevalence of overweight and obesity at one year of age, in the intervention group compared to the control group.

METHODS:

Eleven primary paediatricians randomized to the intervention group and intensively trained about the trial intervention, were asked to consecutively recruit the parents of at least 30 newborns taken in charge within the first six months of the study, and to provide them with standardized oral and written information on protective practices during all the well visits scheduled in the first two years of the child's life. In particular, according to the intervention protocol, parents were provided with oral and written information on behaviors to adopt for their child to be protected from obesity: breast feeding, feeding on demand, responsive feeding, correct time of introduction of complementary feeding, portions shaped on the child's appetite, avoiding "pressing the child to eat more" and rewarding or punishing the child with food, avoiding added sugar and beverages other than milk and water, practicing active game with the child, alternating protein sources correctly and avoiding protein excess. Written menus examples and coloured photos of average portions were given for complementary feeding. Parents were also provided with information about health consequences of childhood obesity.

Another eleven primary paediatricians were randomized to the control group, and asked to consecutively recruit the parents of at least 30 newborns taken in charge within the six months of the study and to provide them with usual care and follow-up.

When all recruited children completed the second year of life, the two groups of toddlers were compared as regards the prevalence of overweight/obesity, defined by WHO cut-offs of the weight/length ratio.

Statistics:

Arm size calculation: although each arm was recruited and followed-up by eleven paediatricians, the minimal number of newborns for each arm was calculated as for a non clustered trial, based on the assumption of a very low intra-class correlation among the newborns recruited by each single paediatrician. Minimal sample size of each arm was calculated in order to have an 80% power to detect, with 95% of statistical certitude, a 33% reduction of overweight/obesity at 24 months of age in the intervention compared to the control arm. This corresponds to about a 18% and a 27% prevalence in the intervention and control arm, respectively, based on epidemiological data from the Northern Italy (Obesity 2006; 14(5):765-9.). The calculation was performed with G power software (http://www.gpower.hhu.de/) and resulted in a minimal number of 330 newborns per arm, which is the reason why each of the eleven paediatricians participating in either arm was asked to recruit at least 30 newborns.

Statistical analyses: rates of overweight/obesity were compared across the two arms by Chi Squared test. Moreover, a binary logistic model was run, with overweight/obesity as dependent variable and arm, parental BMI and parental socio-economic status as independent variables.

The same type of analysis was performed for secondary binary outcomes (rate of overweight/obesity at one year of age, rate of beverage consumption, etc...).

Continuous variables (BMI, weight/lenght ratio) were compared across the two arms by general linear models, with arms as fixed factor and parental BMI and socio-economic status as co-variates.

ELIGIBILITY:
Inclusion Criteria:

Gestational age: 37-42 weeks; no perinatal complication; informed consent from parents.

Exclusion Criteria:

Any congenital disorder, disease or syndrome.

Ages: 5 Days to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 569 (Actual)
Dates: Start 2014-07-01 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Body mass index (BMI) at two years of age. | Third year of the study.
  Overweight = BMI above 85° percentile of the CDC curves; Obesity = BMI above 95° percentile of the CDC curves.

SECONDARY OUTCOMES:
Weight/length ratio at one year of age. | Second year of the study.
  Overweight = ratio above the 85° percentile in the WHO curves.
Beverages at two years of age. | Third year of the study.
  Parents are asked if they usually give their child beverages other than milk or water. (possible answer: yes or no).

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Diabetes and Metabolic Disorders Unit, Department of Life and Reproduction Sciences, University of Verona, 1 Piazzale Stefani, Verona, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pigeot I, Barba G, Chadjigeorgiou C, de Henauw S, Kourides Y, Lissner L, Marild S, Pohlabeln H, Russo P, Tornaritis M, Veidebaum T, Wawro N, Siani A. Prevalence and determinants of childhood overweight and obesity in European countries: pooled analysis of the existing surveys within the IDEFICS Consortium. Int J Obes (Lond). 2009 Oct;33(10):1103-10. doi: 10.1038/ijo.2009.142. Epub 2009 Jul 28. PMID 19636314
- [Background] Reilly JJ, Kelly J. Long-term impact of overweight and obesity in childhood and adolescence on morbidity and premature mortality in adulthood: systematic review. Int J Obes (Lond). 2011 Jul;35(7):891-8. doi: 10.1038/ijo.2010.222. Epub 2010 Oct 26. PMID 20975725
- [Background] Binkin N, Fontana G, Lamberti A, Cattaneo C, Baglio G, Perra A, Spinelli A. A national survey of the prevalence of childhood overweight and obesity in Italy. Obes Rev. 2010 Jan;11(1):2-10. doi: 10.1111/j.1467-789X.2009.00650.x. Epub 2009 Sep 17. PMID 19761508
- [Background] Oude Luttikhuis H, Baur L, Jansen H, Shrewsbury VA, O'Malley C, Stolk RP, Summerbell CD. Interventions for treating obesity in children. Cochrane Database Syst Rev. 2009 Jan 21;(1):CD001872. doi: 10.1002/14651858.CD001872.pub2. PMID 19160202
- [Background] Waters E, de Silva-Sanigorski A, Hall BJ, Brown T, Campbell KJ, Gao Y, Armstrong R, Prosser L, Summerbell CD. Interventions for preventing obesity in children. Cochrane Database Syst Rev. 2011 Dec 7;(12):CD001871. doi: 10.1002/14651858.CD001871.pub3. PMID 22161367
- [Background] Stocks T, Renders CM, Bulk-Bunschoten AM, Hirasing RA, van Buuren S, Seidell JC. Body size and growth in 0- to 4-year-old children and the relation to body size in primary school age. Obes Rev. 2011 Aug;12(8):637-52. doi: 10.1111/j.1467-789X.2011.00869.x. Epub 2011 Mar 23. PMID 21426479
- [Background] Wojcicki JM, Heyman MB. Let's Move--childhood obesity prevention from pregnancy and infancy onward. N Engl J Med. 2010 Apr 22;362(16):1457-9. doi: 10.1056/NEJMp1001857. Epub 2010 Apr 14. No abstract available. PMID 20393165
- [Background] Daniels LA, Mallan KM, Battistutta D, Nicholson JM, Perry R, Magarey A. Evaluation of an intervention to promote protective infant feeding practices to prevent childhood obesity: outcomes of the NOURISH RCT at 14 months of age and 6 months post the first of two intervention modules. Int J Obes (Lond). 2012 Oct;36(10):1292-8. doi: 10.1038/ijo.2012.96. Epub 2012 Jun 19. PMID 22710926
- [Background] WHO Multicentre Growth Reference Study Group. WHO Child Growth Standards based on length/height, weight and age. Acta Paediatr Suppl. 2006 Apr;450:76-85. doi: 10.1111/j.1651-2227.2006.tb02378.x. PMID 16817681
- [Derived] Morandi A, Tommasi M, Soffiati F, Destro F, Fontana L, Grando F, Simonetti G, Bucolo C, Alberti E, Baraldi L, Chiriaco A, Ferrarese N, Frignani G, Pasqualini M, Rossi V, Siciliano C, Zuccolo AM, Matticchio G, Vettori V, Danieli D, Guarda L, Iuliano M, Raimo F, Sirpresi S, Trevisan E, Vinco S, Maffeis C. Prevention of obesity in toddlers (PROBIT): a randomised clinical trial of responsive feeding promotion from birth to 24 months. Int J Obes (Lond). 2019 Oct;43(10):1961-1966. doi: 10.1038/s41366-019-0406-0. Epub 2019 Jul 3. PMID 31270429